CLINICAL TRIAL: NCT02879331
Title: Clinical Study to Evaluate the Exercise Capacity in Patients With Severe Emphysema Treated With Coils
Acronym: CYCLONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC 33-16/IIS-FJD
Record Dates: First submitted 2016-07-29; First posted 2016-08-25 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Emphysema
Keywords: pulmonary emphysema; coils; cycloergometry; lung volume reduction
MeSH Terms: conditions — Pulmonary Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 coils in upper lobes (Active Comparator): 10 coils in upper lobes
  Interventions: Procedure: 10 coils in upper lobes; Procedure: cycloergometry
- 15 coils in upper and lower lobes (Experimental): 15 coils in upper and lower lobes
  Interventions: Procedure: 15 coils in upper and lower lobes; Procedure: cycloergometry

INTERVENTIONS:
Procedure: 10 coils in upper lobes
  Arms: 10 coils in upper lobes
Procedure: 15 coils in upper and lower lobes
  Arms: 15 coils in upper and lower lobes
Procedure: cycloergometry

SUMMARY:
The study hypothesis is that patients with homogeneous emphysema behave differently compared to heterogeneous emphysema with respect to exercise capacity. A better understanding of this difference will allow the investigators to choose the best treatment for each type of patient.

The main purpose of this study is to evaluate the change in exercise capacity measured by cycle ergometry in patients with severe emphysema after endoscopic lung volume reduction with coils (eLVR).

As a secondary purpose, the investigators want to perform an exploratory, randomized study to compare the results of two different therapeutic approaches in a small sample of patients with homogeneous emphysema.

DETAILED DESCRIPTION:
The study plans to include patients with severe emphysema candidates to go through eLVR with coils that fulfill all inclusion criteria and none of the exclusion criteria. Patients with both homogeneous and heterogeneous emphysema will be included.

The main study intervention is the performance of a cyclo ergometry (not included in daily clinical practice) before (basal) and 6 months after going through the eLVR with coils.

The subgroup of patients with homogeneous emphysema will be randomly assigned to the following therapeutic approaches:

* Group A: treatment with 10 coils in upper lobes
* Group B: treatment with 15 coils spared in upper and lower lobes

Thus, the study includes:

* for all patients, the performance of two cycloergometries, before and 6 months after the eLVR
* Also, for the subset of homogeneous emphysema patients, an open label, randomized, parallel, two arm exploratory clinical trial.

Sample size has not been formally calculated as there are no previous available data for the primary endpoint (change inspiratory capacity). Thus, 35 patients will be included according to the expected number of patients. Recruitment period will be 24 months and patient follow up will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Emphysematous patient
* FEV1 < 50%
* RV > 200%
* Diffusion <60% >20%
* PSP <55 mmHg

Exclusion Criteria:

* Anticoagulants/antiplatelets
* Giant bullae (> 8 cm , 1/3 hemithorax)
* More tan three moderate/severe exacerbation per year
* Negative to sign informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Inspiratory Capacity (L) | three months before procedure and six months after first procedure
  Change in Inspiratory Capacity (L) at 6 months from baseline

SECONDARY OUTCOMES:
RV (L) | three months before procedure and six months after first procedure
  Residual Volume (L)
6-MWT (m) | three months before procedure and six months after first procedure
  Six minute walk test (m)
SGQLT (measured in points) | three months before procedure and six months after first procedure
  Saint George quality of life test (points)
FEV1(measured in liters) | three months before procedure and six months after first procedure
  Forced Expiratory Volume in 1 Second (L)
FVC (measured in liters) | three months before procedure and six months after first procedure
  Forced Vital Capacity (L)
Endoscopic Volume Reduction-Associated Complications Rate | 6 months
  Endoscopic Volume Reduction Complications Rate
Cycloergometry-associated Complications Rate | 6 months
  Cycloergometry-associated Complications Rate

CONTACTS AND LOCATIONS:
Overall Officials: Iker Fernandez-Navamuel, MD, PhD, Principal Investigator — FJD
Locations (1):
- Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartman JE, Klooster K, Ten Hacken NH, Slebos DJ. Treatment of emphysema using bronchoscopic lung volume reduction coil technology: an update on efficacy and safety. Ther Adv Respir Dis. 2015 Oct;9(5):251-9. doi: 10.1177/1753465815589904. Epub 2015 Jun 25. PMID 26113524
- [Background] Deslee G, Klooster K, Hetzel M, Stanzel F, Kessler R, Marquette CH, Witt C, Blaas S, Gesierich W, Herth FJ, Hetzel J, van Rikxoort EM, Slebos DJ. Lung volume reduction coil treatment for patients with severe emphysema: a European multicentre trial. Thorax. 2014 Nov;69(11):980-6. doi: 10.1136/thoraxjnl-2014-205221. Epub 2014 Jun 2. PMID 24891327
- [Background] Boutou AK, Zoumot Z, Nair A, Davey C, Hansell DM, Jamurtas A, Polkey MI, Hopkinson NS. The Impact of Homogeneous Versus Heterogeneous Emphysema on Dynamic Hyperinflation in Patients With Severe COPD Assessed for Lung Volume Reduction. COPD. 2015;12(6):598-605. doi: 10.3109/15412555.2015.1020149. Epub 2015 Sep 23. PMID 26398112
- [Background] Aros F, Boraita A, Alegria E, Alonso AM, Bardaji A, Lamiel R, Luengo E, Rabadan M, Alijarde M, Aznar J, Bano A, Cabanero M, Calderon C, Camprubi M, Candell J, Crespo M, de la Morena G, Fernandez A, Ferrero JA, Gayan R, Bolao IG, Hernandez M, Maceira A, Marin E, Muela de Lara A, Placer L, San Roman JA, Serratosa L, Sosa V, Subirana MT, Wilke M. [Guidelines of the Spanish Society of Cardiology for clinical practice in exercise testing]. Rev Esp Cardiol. 2000 Aug;53(8):1063-94. Spanish. PMID 10956604